CLINICAL TRIAL: NCT04840589
Title: Phase I/Ib Trial Evaluating the Safety and Efficacy of BET Inhibitor, ZEN003694 With PD-1 Inhibitor, Nivolumab With or Without CTLA-4 Inhibitor, Ipilimumab in Solid Tumors
Brief Title: Testing the Combination of ZEN003694 and Nivolumab With or Without Ipilimumab in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-02850; NCI-2021-02850 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCC#21-211; 10433 (Other: UPMC Hillman Cancer Center LAO); 10433 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Recurrent Platinum-Resistant Ovarian Carcinoma; Refractory Ovarian Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms | interventions — Biopsy; Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Doublet treatment (ZEN003694, nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and ZEN003694 PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI, a CT scan, a PET scan, and/or an x-ray as well as blood sample collection throughout the trial. Patients also undergo a biopsy during screening.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Procedure: X-Ray Imaging
- Triplet treatment (nivolumab, ZEN003694, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1, ipilimumab IV over 90 minutes on day 1, and ZEN003694 PO QD on days 1-21 or 1-28 of each cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 5, patients are no longer treated with ipilimumab, but receive nivolumab IV over 30 minutes on day 1 and ZEN003694 PO QD on days 1-21 or 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI, a CT scan, a PET scan, and/or an x-ray as well as blood sample collection throughout the trial. Patients also undergo a biopsy during screening and on study.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Procedure: X-Ray Imaging

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Procedure: Biopsy Procedure — Undergo a biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Triplet treatment (nivolumab, ZEN003694, ipilimumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo a PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I/Ib trial is to find out the best dose, possible benefits and/or side effects of BET bromodomain inhibitor ZEN-3694 (ZEN003694) when given in combination with nivolumab with or without ipilimumab in treating patients with solid tumors. ZEN003694 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving ZEN003694 in combination with nivolumab with or without ipilimumab may shrink or stabilize solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety/tolerability and recommended phase 2 dose (RP2D) of the BET inhibitor (BETi) ZEN003694 when combined with nivolumab with or without low dose ipilimumab in solid tumors.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the triplet regimen in a cohort of patients with recurrent platinum-resistant BRCA wild type (wt) epithelial ovarian cancer.

Ia. To observe and record anti-tumor activity. II. To evaluate the impact of BET inhibition on the tumor immune microenvironment (TIME).

III. To explore predictors of response and resistance to therapy. IV. To characterize the pharmacokinetic (PK) profile of ZEN003694 and its active metabolite ZEN003791.

EXPLORATORY OBJECTIVE:

I. To correlate drug exposure with response and/or toxicity.

OUTLINE: This is a dose-escalation study of ZEN003694 followed by a dose-expansion study.

DOSE ESCALATION (DOUBLET TREATMENT): Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and ZEN003694 orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI), a computed tomography (CT) scan, a positron emission tomography (PET) scan, and/or an x-ray as well as blood sample collection throughout the trial. Patients also undergo a biopsy during screening.

DOES ESCALATION AND DOSE EXPANSION (TRIPLET TREATMENT): Patients receive nivolumab IV over 30 minutes on day 1, ipilimumab IV over 90 minutes on day 1, and ZEN003694 PO QD on days 1-21 or 1-28 of each cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 5, patients are no longer treated with ipilimumab, but receive nivolumab IV over 30 minutes on day 1 and ZEN003694 PO QD on days 1-21 or 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI, a CT scan, a PET scan, and/or an x-ray as well as blood sample collection throughout the trial. Patients also undergo a biopsy during screening and on study.

After completion of study treatment, patients are followed up for 30 days, then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic or recurrent solid tumor malignancy for which standard curative or palliative measures do not exist or are no longer effective

  * Dose escalation/phase I: Metastatic or recurrent solid tumors with measurable or evaluable disease
  * Dose expansion exploratory cohorts (nivolumab + ipilimumab + ZEN003694): Recurrent BRCAwt epithelial ovarian carcinoma patients who have progressed or recurred within < 6 months from prior platinum-based therapy
* Dose escalation and expansion exploratory cohorts: Patients must have measurable and biopsiable disease (at least two lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. For patients in the dose escalation with evaluable disease, biopsy is mandated if feasible
* No more than 5 lines of prior therapy for the dose escalation and expansion phases

  * In the expansion cohorts, up to 2 prior lines in the platinum-resistant setting is allowed
  * Patients with primary refractory ovarian cancer (who progressed while on primary 1L platinum therapy) will be excluded in the dose expansion cohorts but allowed in the dose escalation cohort
* Patients who have had chemotherapy or radiotherapy more than 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study and who have recovered from adverse events due to agents administered more than 4 weeks earlier are eligible; for oral therapies, a patient is eligible after 5 half-lives of the drug. Prior palliative (limited field) radiation therapy is permitted, if all of the following criteria are met:

  * Palliative radiation must have been completed at least 4 weeks before starting study treatment
  * Repeat imaging demonstrates no new sites of bone metastases
  * Irradiated sites of metastasis should not be selected as target lesions
  * Patients must have recovered to meet all eligibility criteria
* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of nivolumab in combination with ZEN003694 +/- ipilimumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 150,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine clearance (CrCl) >= 60 mL/min (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better and have a corrected QT (QTc) interval < 450 msec
* The effects of nivolumab, ZEN003694, and/or ipilimumab on the developing human fetus are unknown. For this reason and because nivolumab, ZEN003694, and/or ipilimumab are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of investigational drug. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception.

  * WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
  * WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of investigational product. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days.
  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients with sarcoma or non-epithelial histology
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to the first dose of study intervention
* Prior therapy with PD-1, PD-L1, or CTLA-4 inhibitors, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways. Prior anti-PD-1/PD-L1 in microsatellite instability-high (MSI-H) tumors is allowed in the dose escalation cohort if no grade 2 or more toxicities developed during that therapy requiring stopping immune checkpoint inhibition. Patients who have received prior vaccine therapy are eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, ipilimumab, and/or ZEN003694, including severe hypersensitivity reactions to any monoclonal antibody
* Patients who are receiving any other investigational agents
* Patients with human immunodeficiency virus (HIV) infection may be enrolled on this study provided: (a) they are on a stable regimen of highly active anti-retroviral therapy (HAART) with no medications otherwise prohibited by this protocol (e.g. drug-drug interactions,), e.g. medications cannot be CYP3A4 inducers or inhibitors and cannot interact with ZEN003694), and (b) they require no concurrent antibiotics or antifungals for the prevention of opportunistic infections, and (c) they have a CD4 count above 250 cell/mcL and an undetectable viral load on standard polymerase chain reaction (PCR)-based tests within 1 month of initiation of study treatment
* Other patients with clinically significant immunosuppression, e.g. organ transplant patients, are not eligible. If clarification is needed, this may be discussed with the medical monitor. Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection. Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* Patients with known immune impairment who may be unable to respond to anti-CTLA-4 antibody
* Bowel obstruction or any condition precluding oral intake. No gastric tube for venting purposes. No significant gastrointestinal disease or fistula
* Known active hepatitis infections or active infections require IV systemic antibiotics
* Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 or that receive fluoxetine (moderate CYP2C19 inhibitor with a metabolite that potentially causes CYP3A4 inhibition) are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association Classification class II), or serious cardiac arrhythmia requiring medication
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* Pregnant women are excluded from this study because nivolumab and ipilimumab are immunotherapeutic agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab and ipilimumab, breastfeeding should be discontinued if the mother is treated with nivolumab and ipilimumab. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 1 cycle of treatment for doublet group (4 weeks) and up to 2 cycles for triplet group (6 weeks)
  Will calculate maximum tolerated dose and dose limiting toxicity with dose escalation using standard 3+3 design.
Phase 2 recommended dose for the combined regimens | Up to 1 cycle of treatment for doublet group (4 weeks) and up to 2 cycles for triplet group (6 weeks)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year post-treatment
  Defined as partial or complete response to the combined regimens in the entire cohort and in the expansion cohort. Assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) only. All treatment decisions should be made by RECIST v1.1 only.
Progression-free survival | Up to 1 year post-treatment
Overall survival | Up to 1 year post-treatment
Incidence of adverse events | Up to 1 year post-treatment
  Will include grade 3 and 4 immune and non-immune events assessed by Common Terminology Criteria for Adverse Events version 5.0.
Clinical benefit | Up to 1 year post-treatment
  Defined as ORR and stable disease.
Whole exome sequencing | Up to 1 year post-treatment
  Will assess: a) CCNE1, MYC, BRD4 status b) MSI status and tumor mutational burden c) B2M mutation/deficiency and alteration in antigen processing/presentation machinery (MHC1) d) Alteration in other molecular pathways such as HRD/BRCA, PI3K.
Next generation sequencing ribonucleic acid sequencing | Up to 1 year post-treatment
  Will assess: a) Functional CCNE1, MYC, BRD4 gene expression status at baseline and at 4 weeks b) Alteration in tumor immune microenvironment and immune markers/signature like interferon-gamma signature.
PD-L1 expression in tumor cells and tumor-associated immune cells | Up to 1 year post-treatment
Multiplex analysis of tumor infiltrating immune cells | Up to 1 year post-treatment
  Will assess immune cell subpopulations and their activation status.
Pharmacokinetic (PK) parameters | Pre dose, and then 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 h after dose on cycle 1, day 1; and pre dose and 1-3 hours post-dose on cycle 2, day 1
  Individual PK parameters will be estimated, specifically maximum concentration, area under the concentration-time curve, half-life, apparent clearance, and apparent volume of distribution using non-compartmental methods. The PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. PK parameters will be reported descriptively for exploratory comparison with historical data.
Phenotypic characteristics of peripheral blood mononuclear cells over treatment | At 4 weeks (cycle 2 day 1 of treatment)
  Will compare these phenotypic characteristics to baseline to assess different immune cells subset and their activation status peripherally.
Circulating tumor deoxyribonucleic acid | Up to 1 year post-treatment
  Assessed in plasma using TSO500 panel. Will assess: a) CCNE1, MYC, and BRD4 (if BRD4 became available) status at baseline and during treatment to assess if blood-based status is concordant with tissue based status and if the status changes during therapy b) Blood based molecular residual disease and tumor mutational burden.
Pro-inflammatory and anti-inflammatory cytokines analyses | Up to 1 year post-treatment
  Assessed in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Haider S Mahdi, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (9):
- United States (9):
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Feng Y, Mahdi H, Piekarz R, Beumer JH, Synold TW. An LC-MS/MS method for determination of the bromodomain inhibitor ZEN-3694 and its metabolite ZEN-3791 in human plasma. Bioanalysis. 2024;16(8):227-238. doi: 10.4155/bio-2023-0252. Epub 2024 Mar 18. PMID 38497709